CLINICAL TRIAL: NCT04230915
Title: Low-dose Rocuronium Provides Adequate Muscle Relaxation and Increases the Effectiveness of Intraoperative Neural Monitoring in Thyroid Surgery
Brief Title: Low-dose Rocuronium Effect Neural Monitoring in Thyroid Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BakirkoySadiKonuk -2019/154
Record Dates: First submitted 2019-11-25; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Thyroid
Keywords: Intraoperative nerve monitoring; Train of four (TOF); Rocuronium; Operation Time
MeSH Terms: conditions — Thyroid Diseases | interventions — Intraoperative Neurophysiological Monitoring

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Dose Rocuronium (Active Comparator): This group patients will determine as those who were administered 0.3 mg/kg rocuronium
  Interventions: Other: Intraoperative nerve monitoring
- Strandart Dose Rocuronium (No Intervention): This group patients will determine as those who were administered 0.6 mg/kg rocuronium

INTERVENTIONS:
Other: Intraoperative nerve monitoring — This group will determine as those who were administered 0.3 mg/kg rocuronium,
  Arms: Low Dose Rocuronium

SUMMARY:
Intraoperative Neuromonitoring (IONM) was started to be used by surgeons to help prevent laryngeal nerve (RLN) damage during thyroid and parathyroid operations. IONM can be used to localize and identify RLN intraoperatively, to evaluate vocal function after thyroid resection, and to explain the mechanism of RLN injury. However, an important problem in the routine use of IONM is the effect of neuromuscular blocking agents (NMBAs). The use of NMBAs in general anesthesia is essential to provide clinically acceptable tracheal intubation conditions and to prevent laryngeal trauma. However, NMBAs may be the potential cause of a false-negative response during the IONM. Randolph et al. proposed short-acting 1-2 mg/kg succinylcholine for enough relaxation and the ease of electromyographic (EMG) endotracheal tube intubation during the IONM. However, succinylcholine, a depolarizing NMBA, is associated with various adverse effects such as cardiac arrhythmia, hyperkalemia, and malignant hyperthermia. Nondepolarizing NMBAs are widely used by most anesthesiologists due to their safe effects, but to the best our knowledge, there is no very short-acting nondepolarizing NMBA. This deficiency creates a problem because the dose and the time point of nerve stimulation are critical for a successful IONM. However, some studies have reported the feasibility of IONM following the administration of nondepolarizing NMBAs during a thyroid operation. Rocuronium is a short-acting and nondepolarizing NMBA type which is widely used for induction in general anesthesia. Although 0.6 mg/kg rocuronium is recommended for standard intubation dose, the ease of intubation can also be provided with 0.3 mg/kg rocuronium or 1.5 mg/kg succinylcholine. Therefore, the present study was designed to compare the effects of IONM with low and standard rocuronium doses in the induction of general anesthesia.

DETAILED DESCRIPTION:
The present study was approved by the local Institutional Review Board. A written informed consent form was obtained from each patient. Patients were informed on the purpose of using the INOM system to potentially assist in the localization and identification of RLNS during the operation as well as to evaluate their functions.

The study includes patients between the ages of 18-65 who were implemented total thyroidectomy, those with ASA I-III, patients who were approved by the otolaryngologist to have a normal cord examination before and after surgery and patients operated by 2 surgeons who were general surgery specialists and accepted as endocrine surgery consultants and anesthetized by the only anesthesiologist who was included in the study.

The exclusion criteria were determined as predicted difficult intubation, severe liver or renal dysfunction, asthma, drug abuse, morbid obesity, and the presence of drug use that may affect neuromuscular diseases or neuromuscular transmissions.

The study was designed as a prospective randomized controlled and double-blind study. Accidental numbers were produced in order to prevent selection bias. In the numbers produced, 1: 0,3 mg/kg rocuronium, 2: 0,6 mg/kg rocuronium group was predefined and patients were assigned to groups in this direction. Random numbers made MedCalc 18.2.1. The double-blind study was designed in a way that the anesthesia technician who gave the rocuronium to the anesthesiologist knew, and the anesthesiologist and surgeon who intubated and carried out the TOF and INOM follow-up didn't know the groups.

The group 1 patients were determined as those who were administered 0.3 mg/kg rocuronium, and the group 2 patients as those who were administered 0.6 mg/kg rocuronium.

For the patients who were taken to the operation table, EKG, SPO2, TA, TOF monitorization will be performed and the values will be recorded during the operation. The anesthesia induction of both groups will be done with 3 mg/kg propofol, 2 mg/kg fentanyl and rocuronium bromide according to the relevant group and an intubation tube with the appropriate number and having the IONM electrode will be used as intubation tube for each patient (NIM).

The neuromuscular blockade was followed up quantitatively with an acceleromiograph (TOF Guard; Organon Teknika NV, Turnhout, Belgium). The stimulation of the ulnar nerve and acceleration measurements for the adductor pollicis muscle were used for the acceleromiography. Electrodes were placed on the ulnar nerve at the volar surface of the wrist. The distal electrode was placed at the point where the proximal bending line passed to the radial side of the flexor carpi ulnaris muscle.

The proximal electrode was placed 2 or 3 cm proximally on the distal electrode. The converter (TOF-Watch Handadapter; Organon) was positioned in a way that the largest flat surface corresponds to the thumb. The converting cable was placed so that no traction was applied to the converter and the movement of the thumb was not restricted in any way.

Following the anesthesia induction, rocuronium was administered to the group at an appropriate dosage and the patients who had a TOF value below 90% were intubated. The EMG endotracheal tube (Nerve Integrity Monitor [NIM]; Medtronic Xomed, Jacksonville, FL) was placed directly by an anesthesiologist with laryngoscopy. The position of the electrodes was checked by a laryngoscopic examination after the patient's neck was placed in the full extension position according to our standard IONM procedures.

The anesthesia maintenance after induction was achieved with 2-3% severane and 0.05-0.2 micgr / kg remifentanil. A 40 mg-propofol was added as the recovery dose during the surgery.

Vagal stimulation is the routine procedure prior to the definition of RLN during thyroid operation. This step is important to ensure that the monitoring system is working correctly and that the RLN remains on a normal path. The vagus nerve was found first when the skin flap was removed.

The nerve was then stimulated every 5 min after 30 to 70 minutes following the administration of the rocuronium. 8 EMG signals were measured at 30th, 35th, 40th, 45th, 50th, 55th, 60th, and 70th minutes, respectively. To obtain an EMG response, the vagus nerve was directly touched with a 2 mA monopolar nerve stimulus bar (Prass; Medtronic Xomed).

The Helbo-Hansen score (Steyn's modification, Table1) was used to evaluate the ease of intubation. The sum of the scores of these five individual variables was calculated as the Helbo-Hansen score (Steyn's modification, Table 1). A total score of 5 points was considered to be excellent, 6-10 points to be good, 11-15 points to be bad, and 16-20 points to be too bad.

The statistical analysis of continuous variables between groups was compared using 2 samples t-tests. The intra-group statistical analyses of continuous variables were compared by using the paired t-test. The categorical nominal variables were analyzed by the chi-square test or Fisher's exact test. All statistical tests were 2-tailed and the probability of p<0.05 was considered as statistically significant. All data were expressed as mean ± standard deviation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis of nodular or multinodular goiter
* Clinical, radiological and pathologicllay diagnosed thyroid cancer
* Must be able to speak( for voice recording)

Exclusion Criteria:

* Pregnancy
* Previous thyroid surgery
* Previous laryngeal surgery
* Professional voice users( e.g. singers)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-04-29 (Estimated); Study Completion 2020-04-29 (Estimated)

PRIMARY OUTCOMES:
Nerve signal detection time | Duration of surgery, up to 3 hours
  Variation of nerve signal detection time with dose of rocuronium

SECONDARY OUTCOMES:
Operation time | Duration of surgery, up to 3 hours
  Comparison of differences in operation time period between the groups whether IONM

CONTACTS AND LOCATIONS:
Locations (1):
- Bakırkoy Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)